CLINICAL TRIAL: NCT00620529
Title: A Clinical Trial to Measure the Effect of DHA-enriched Fish Oils on Blood Pressure, Heart Rate Variability and Liver Fat Content in the Polycystic Ovary Syndrome
Brief Title: The Effects of Fish Oils on Blood Pressure, Heart Rate Variability and Liver Fat in the Polycystic Ovary Syndrome
Acronym: fops
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keogh Institute for Medical Research (Other)
Collaborators: Royal Perth Hospital (Other)
Responsible Party: Dr Andrea Cussons, University of Western Australia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC 2008/049
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; cardiovascular risk; metabolism; blood pressure; liver fat; heart rate variability
MeSH Terms: conditions — Polycystic Ovary Syndrome; Fatty Liver | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 20/50 fish oil, 1000mg capsules, Ocean Nutrition 2050,4g/day.
  Interventions: Dietary Supplement: Ocean Nutrition 2050
- 2 (Placebo Comparator): olive oil capsules
  Interventions: Dietary Supplement: Olive oil capsules

INTERVENTIONS:
Dietary Supplement: Ocean Nutrition 2050 — 1000mg capsules, 4 capsules/day for 8 weeks
  Other Names: Code name: 2050
  Arms: 1
Dietary Supplement: Olive oil capsules — Olive oil capsules, 4 per day for 8 weeks
  Arms: 2

SUMMARY:
We hypothesise that fish oils will have a beneficial effect on cardiometabolic parameters in women with PCOS. The purpose of this study therefore is to examine the effects of fish oils on blood pressure, heart rate variability and liver fat content in obese women with the polycystic ovary syndrome.

DETAILED DESCRIPTION:
The prevalence of abnormalities of blood pressure (ABP), variability of heart rate (HRV) and liver fat content is increased in women with the polycystic ovary syndrome (PCOS). We hypothesise that fish oils will have a beneficial effect on these endpoints and other cardiometabolic parameters such as cholesterol and liver function in women with PCOS. This crossover study of 40 obese women with PCOS will therefore examine the effects of fish oils on the above parameters compared with placebo (olive oil). Subjects with PCOS who have participated in previous studies with this research group will be approached for recruitment, as will eligible subjects within the endocrine clinics of the chief and co-investigators.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese women with PCOS as per 1990 NIH criteria (see below)
* Non-smokers
* Age>18 years, premenopausal
* Acceptable to have/be on treatment for type 2 diabetes mellitus and/or dyslipidaemia
* Acceptable to be taking the oral contraceptive pill

Exclusion Criteria:

* Uncontrolled hypertension (BP>160/100mmHg)
* Known co-morbidities including liver or renal disease
* Already taking fish oil supplements
* Other intercurrent illness (major surgery, CV event)
* Smokers
* Alcohol intake >20g/day
* Pregnancy
* Any metallic implant (contraindication for MRI).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
24 hour ambulatory systolic blood pressure | week 8 and week 24

SECONDARY OUTCOMES:
24 hour heart rate variability | week 8 and week 24
liver fat content (MRI) | week 8 and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Andrea J Cussons, MBBS, Principal Investigator — The University of Western Australia
Locations (1):
- School of Medicine and Pharmacology, Royal Perth Hospital, Perth, Western Australia, Australia